CLINICAL TRIAL: NCT06594250
Title: Study of the Nasal Intracellular Reservoir of Staphylococcus Aureus in Patients With S. Aureus Bacteremia
Acronym: RISTA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH025; 2020-A02692-37 (Other: ANSM)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bacteria Infection Mechanism
Keywords: Staphylococcus aureus bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We plan to conduct a study to assess the frequency of the intracellular S. aureus reservoir (within carriers) in S. aureus bacteremia and in bacteremia to another pathogen (control group). We would also like to study the impact of this reservoir on the persistence of carriage and prognosis (death, duration of bacteremia, length of stay, presence of secondary localizations of bacteremia or endocarditis in the case of S. aureus bacteremia).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Experimental group comprising patients with S. aureus bacteremia with or without IE
  Interventions: Diagnostic Test: Nasal swab; Biological: Venous sampling; Biological: Antibiotic treatment; Device: Nasal swab; Biological: Intracellular reservoir test
- Control group: Control group comprising patients with bacteremia with a pathogenic bacterial species other than S. aureus with or without IE.
  Interventions: Diagnostic Test: Nasal swab; Biological: Venous sampling; Biological: Antibiotic treatment; Device: Nasal swab; Biological: Intracellular reservoir test

INTERVENTIONS:
Diagnostic Test: Nasal swab — Nasal swab to detect nasal carriage of S. aureus
Biological: Venous sampling — Peripheral venous sampling to collect peripheral blood mononuclear cells.
Biological: Antibiotic treatment — Antibiotic treatment for bacteremia (+/- 1 month), in all patients with S. aureus
Device: Nasal swab — A new nasal swab will be taken using the same technique, to see whether or not the carriage persists
Biological: Intracellular reservoir test — In the event of positive carriage, a new intracellular reservoir test will be performed. A search for relapse (new S. aureus infection) or recurrence (S. aureus bacteremia if the 1st bacteremia was due to another pathogen) will be carried out.

SUMMARY:
Staphylococcus aureus bacteremia is a serious infection associated with a high mortality rate (with or without associated infective endocarditis (IE)), long hospital stays and multiple complications, due to the terrain in which it occurs and its secondary localization. They may be community-acquired or healthcare-associated infections. Being a carrier of S. aureus is a known risk factor for S. aureus bacteremia. Although several mucosal sites of carriage have been described, screening for carriage is most often carried out at the nasal level, both for reasons of simplicity and because it is the predominant site of carriage of this bacterium. However, S. aureus carriage is a frequent occurrence, affecting around 1/3 of the general population.

DETAILED DESCRIPTION:
Long considered an extracellular bacterium, the investigators now know that S. aureus can have an intracellular reservoir. This was initially described in situations of infection (bone infections, vascular infections) and more recently in situations of nasal carriage without associated infection. Among S. aureus carriers, between 15% and 30% have an intracellular reservoir of this bacterium, depending on the study, in patients with no S. aureus infection. For S. aureus carriers with S. aureus infection, there are no data in the literature. The clinical significance of this intracellular reservoir in a carrier situation is currently unknown. The study team was able to demonstrate in vitro that this reservoir was not affected by the mupirocin used in decolonization, and preliminary results suggest that in vivo this reservoir may also be associated with decolonization failure.

Moreover, in vitro, it has been suggested that S. aureus may act on autophagy to promote intracellular survival. Is the intracellular reservoir more frequent in patients with S. aureus bacteremia? Is it associated with a poorer prognosis in S. aureus bacteremia? Is it associated with the production of certain S. aureus intracellular persistence factors? Is it associated with a slowdown in autophagic flow in nasal cells or phagocytes? These questions remain unanswered to this day.

To explore these questions, the investigators plan to conduct a study to assess the frequency of the intracellular S. aureus reservoir (within carriers) in S. aureus bacteremia and in bacteremia to another pathogen (control group). They would also like to study the impact of this reservoir on the persistence of carriage and prognosis (death, duration of bacteremia, length of stay, presence of secondary localizations of bacteremia or endocarditis in the case of S. aureus bacteremia).

ELIGIBILITY:
Inclusion Criteria:

* Bacteremia
* Patient affiliated or entitled to a social security plan
* Patient who has signed a consent form to participate in the study.

Exclusion Criteria:

* Antibiotic therapy in place for more than 5 days at the time of inclusion
* Nasal decolonization of S. aureus within 12 months
* Pregnant or breast-feeding women
* Patients under guardianship
* Polymicrobial bacteremia including S. aureus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at St-Etienne University Hospital with bacteremia with or without IE. Patients will be assigned to the experimental group in the case of S. aureus bacteremia (whether or not associated with an IE), or to the control group in the case of bacteremia caused by a pathogenic bacterium other than S. aureus (whether or not associated with an IE).
Sampling Method: Non-Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of intracellular S. aureus carriers at nasal level research | At inclusion
  Number of intracellular S. aureus carriers at nasal level research in patients with S. aureus bacteremia associated or not

SECONDARY OUTCOMES:
Number of intracellular S. aureus carriers at nasal level research | Day 7
In-hospital mortality rate (%) | Month 1
  In-hospital mortality rate directly related to infection (septic shock, multivisceral failure, death during surgical management related to infection) during bacteremia
Mean duration of S. aureus bacteremia (Day) | Month 1
Average number of secondary localizations of S. aureus bacteremia | Month 2
  Clinically diagnosed, or on examination carried out as part of the extension work-up performed as part patient management (Scan, echocardiography, scintigraphy, etc.)
Average length of stay in hospital for S. aureus bacteremia (Day) | Month 1
Proportion of nasal S. aureus carriers still carriers at the end of treatment for bacteremia (%) | Month 1
Proportion of nasal S. aureus carriers still carriers one year after the end of treatment for bacteremia (%) | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth BOTELHO-NEVERS, MD-PhD, Principal Investigator — CHU SAINT-ETIENNE; Léo SAUVAT, MD, Study Chair — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de St Etienne, Saint-Etienne, France